CLINICAL TRIAL: NCT01939717
Title: A Randomized Controlled Pilot Trial Comparing Irish Set Dancing to Usual Care for People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, Joanne Shanahan, Joanne Shanahan, B.S.c, MISCP, University of Limerick
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ST2
Record Dates: First submitted 2013-08-25; First posted 2013-09-11 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Irish set dancing
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dance group (Other): Participants allocated to this group will continue with their usual care and participate in a set dancing class.
  Interventions: Other: Dance group
- Control group (No Intervention): Participants allocated to this group will act as a control group and continue to receive their usual care only.

INTERVENTIONS:
Other: Dance group — Participants will attend ten weeks of set dancing classes. Each class will be one and half hours. Family members will be invited to partner each participant with Parkinson's disease during the class. Set dancing steps and sets will be thought and progressed in line with the participants abilities. Frequent rests will be taken during the classes.
  Participants will be given a home exercise programme which will involve chair based exercises, mental rehearsal, listening music, watching a dance DVD and practicing dance material thought in class.
  Arms: Dance group

SUMMARY:
Primary aim is to conduct a pilot trial to determine:

1. The feasibility and efficiency of randomisation procedures and study design
2. If recruitment rates are sufficient to adequately power a larger trial

The secondary aim is to determine the efficiency of set dancing in comparison to a control for people with Patkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of idiopathic Parkinson's disease (Hackney et al 2007; Marchant et al 2010), stage 1-2.5 on the modified Hoeln and Yahr scale for staging of Parkinson's disease (Batson 2010)
* Able to walk three meters with an assistive device
* Over 18 years of age
* Not pregnant
* Have access to a computer/DVD player to allow them to participate in the home exercise programme

Exclusion Criteria:

* A serious cardiovascular and/or pulmonary condition (Lodder et al 2004)
* A neurological deficit other than Parkinson's disease (Batson 2010; Marchant et al 2010)
* Evidence of a musculoskeletal problem (Duncan and Earhart 2012), contraindicating participation in exercise participation(Lodder et al 2004)
* A cognitive or hearing problem which will affect their ability to follow instructions or hear the music (Batson 2010)
* Participated in regular dance classes in the past six months (Marchant et al 2010)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of randomization procedures (To assess implementation of randomization procedures) | This outcome measure will be assessed over a 1 year period from study inception to completion
Attrition (To assess dropout rate during the study) | This outcome measure will be assessed over a 1 year period from study inception to completion
  Attrition rate of ≤ 20% per group will be deemed acceptable
Intervention adherence (To assess compliance with the dance intervention) | This outcome will be assessed during the 10 week set dancing intervention
  2) Intervention will be considered successful if no adverse effects or safety issues are reported and attendance at classes is ≥70%
Recruitment rates (To assess rate, duration and success of recruitment methods) | This outcome will be assessed over a one year recruitment period
  Recruitment considered successful and feasible is 100 participants are recruited in one year
Resources (To assess availability of personnel and building needed to implement study methodology) | This outcome measure will be assessed over a 1 year period from study inception to completion
  Document issues regarding availability of personnel or buildings needed to implement study methodology

SECONDARY OUTCOMES:
Exit Questionnaire (To assess participants satisfaction) | This outcome will be assessed the week after the intervention period ends.
  The exit questionnaire will assess participants' satisfaction with the dance intervention at the end of the study. The questionnaire asks participants if they have noted improvements in different aspects of physical well-being, and allows feedback relating to the structure, material and enjoyment of the dance classes to be gathered. This questionnaire has previously been used in other studies investigating the benefit of dance for those with Parkinson's disease (Hackney and Earhart 2009; Hackney and Earhart 2010).
The Parkinson's Disease Questionnaire (PDQ-39) (To assess change in health related quality of life) | This outcome will be assessed within a week before the intervention begins and within a week after the intervention period ends
  Self-report quality of life questionnaire
Unified Parkinson's Disease Rating Scale 3 (UPDRS-3) (To assess changes in motor impairment) | This outcome will be assessed within a week before the intervention begins and within a week after the intervention period ends
  Disease specific measure of motor function
Six minute walk test (To assess change in functional endurnace) | This outcome will be assessed within a week before the intervention begins and within a week after the intervention period ends
  Measure of functional endurance
MiniBESTest (To asses change in balance) | This outcome will be assessed within a week before the intervention begins and within a week after the intervention period ends
  Balance measure

CONTACTS AND LOCATIONS:
Overall Officials: Meg E Morris, Prof., Study Chair — Department of Physiotherapy, School of Allied Health, La Trobe University, Bundoora 3086, Australia.
Locations (1):
- University of Limerick, Limerick, Munster, Ireland

REFERENCES:
- [Background] Duncan RP, Earhart GM. Randomized controlled trial of community-based dancing to modify disease progression in Parkinson disease. Neurorehabil Neural Repair. 2012 Feb;26(2):132-43. doi: 10.1177/1545968311421614. Epub 2011 Sep 29. PMID 21959675
- [Background] Heiberger L, Maurer C, Amtage F, Mendez-Balbuena I, Schulte-Monting J, Hepp-Reymond MC, Kristeva R. Impact of a weekly dance class on the functional mobility and on the quality of life of individuals with Parkinson's disease. Front Aging Neurosci. 2011 Oct 10;3:14. doi: 10.3389/fnagi.2011.00014. eCollection 2011. PMID 22013420
- [Background] Marchant D, Sylvester JL, Earhart GM. Effects of a short duration, high dose contact improvisation dance workshop on Parkinson disease: a pilot study. Complement Ther Med. 2010 Oct;18(5):184-90. doi: 10.1016/j.ctim.2010.07.004. Epub 2010 Aug 21. PMID 21056841
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Shanahan J, Morris ME, Bhriain ON, Volpe D, Lynch T, Clifford AM. Dancing for Parkinson Disease: A Randomized Trial of Irish Set Dancing Compared With Usual Care. Arch Phys Med Rehabil. 2017 Sep;98(9):1744-1751. doi: 10.1016/j.apmr.2017.02.017. Epub 2017 Mar 21. PMID 28336345
- [Derived] Shanahan J, Morris ME, Bhriain ON, Volpe D, Richardson M, Clifford AM. Is Irish set dancing feasible for people with Parkinson's disease in Ireland? Complement Ther Clin Pract. 2015 Feb;21(1):47-51. doi: 10.1016/j.ctcp.2014.12.002. Epub 2014 Dec 13. PMID 25557584